CLINICAL TRIAL: NCT00673205
Title: A Randomized, Double-Blind, Parallel-Group Trial Comparing Bicalutamide (Casodex) 150mg Once Daily With Placebo in Patients With Non-metastatic Prostate Cancer
Brief Title: (Bicalutamide) Casodex vs Placebo in Non-metastatic Early Prostate Cancer
Acronym: Capri
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr. Tom Morris, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D6876C00024; 7054IL/0024
Record Dates: First submitted 2008-05-02; First posted 2008-05-07 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Non-Metastatic Prostate Cancer
Keywords: androgen antagonists; prostate neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator)
  Interventions: Drug: Placebo
- B (Active Comparator)
  Interventions: Drug: Bicalutamide

INTERVENTIONS:
Drug: Bicalutamide — 150mg p.o. daily
  Other Names: Casodex
  Arms: B
Drug: Placebo
  Arms: A

SUMMARY:
The purpose of this trial is to study the effect of adjuvant or immediate hormonal therapy, versus placebo, in subjects who have either undergone a primary therapy (principally radical prostatectomy or radiotherapy) or who were otherwise to be managed by watchful waiting.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of non-metastatic cancer of the prostate gland
* Patient to be 18 years and above

Exclusion Criteria:

* Previous systemic therapy for prostate cancer
* Previous history of another form of cancer (not prostate) within 5 years of study start.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3588 (Actual)
Dates: Start 1995-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Time to clinical progression | Throughout study period
Tolerability in terms of adverse events and laboratory parameters | Throughout study period

SECONDARY OUTCOMES:
Survival | Throughout study period
Time to treatment failure | Throughout study period
Prostate-specific antigen | Initial study period up to 2005 amended protocol

CONTACTS AND LOCATIONS:
Overall Officials: Manfred P Wirth, Professor, Principal Investigator — Technical University of Dresden, Germany
Locations (128):
- Australia (2):
  - Research Site, Wooloongabba, Queensland
  - Research Site, East Melbourne, Victoria
- Austria (5):
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Mistelbach
  - Research Site, Oberwart
  - Research Site, Sankt Pölten
- Belgium (9):
  - Research Site, Antwerp
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Kortrijk
  - Research Site, Leuven
  - Research Site, Mons
  - Research Site, Ostend
  - Research Site, Seraing
- Czechia (4):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- Germany (12):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Dresden
  - Research Site, Freiburg im Breisgau
  - Research Site, Heidelberg
  - Research Site, Jena
  - Research Site, Lübeck
  - Research Site, Lüdenscheid
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Regensburg
  - Research Site, Sigmaringen
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
- Research Site, Dublin, Ireland
- Israel (4):
  - Research Site, Haifa
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (18):
  - Research Site, Bari, BA
  - Research Site, Bergamo, BG
  - Research Site, Belluno, BL
  - Research Site, Bologna, BO
  - Research Site, Brescia, BS
  - Research Site, Como, CO
  - Research Site, Cesena, FO
  - Research Site, Anagni, FR
  - Research Site, Carpi, MO
  - Research Site, Fidenza, PR
  - Research Site, Roma, Roma
  - Research Site, Siena, SI
  - Research Site, Torino, TO
  - Research Site, Treviso, TV
  - Research Site, Udine, UD
  - Research Site, Varese, VA
  - Research Site, Dolo, VE
  - Research Site, Portogruaro, VE
- Research Site, México, Mexico
- Netherlands (13):
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Capelle aan den IJssel
  - Research Site, Eindhoven
  - Research Site, Enschede
  - Research Site, Gouda
  - Research Site, Heerlen
  - Research Site, Maastricht
  - Research Site, Nijmegen
  - Research Site, Roosendaal
  - Research Site, Rotterdam
  - Research Site, Spijkenisse
  - Research Site, Utrecht
- Poland (2):
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Portugal (5):
  - Research Site, Almada
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Vila Nova de Gaia
- South Africa (8):
  - Research Site, Somerset West, Cape Town
  - Research Site, Bloemfontein, South Africa
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, George
  - Research Site, Johannesburg
  - Research Site, Pietermarizberg
  - Research Site, Pretoria
- Spain (18):
  - Research Site, Granada, Andalusia
  - Research Site, Málaga, Andalusia
  - Research Site, Seville, Andalusia
  - Research Site, Bilbao, Basque Country
  - Research Site, Salamanca, Castille and León
  - Research Site, Guadalajara, Castille-La Mancha
  - Research Site, Badalona(barcelona), Catalonia
  - Research Site, Barcelona, Catalonia
  - Research Site, Hospitalet de Llobregat(barcel, Catalonia
  - Research Site, A Coruña, Galicia
  - Research Site, Vigo(pontevedra), Galicia
  - Research Site, Alcalá de Henares, Madrid
  - Research Site, Getafe, Madrid
  - Research Site, Madrid, Madrid
  - Research Site, Pamplona, Navarre
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, San Juan(alicante), Valencia
  - Research Site, Valencia, Valencia
- United Kingdom (23):
  - Research Site, Reading, Berkshire
  - Research Site, Colchester, Essex
  - Research Site, Barnet, Hertfordshire
  - Research Site, Tooting, London
  - Research Site, Belfast, Northern Ireland
  - Research Site, Taunton, Somerset
  - Research Site, Gwent, South Wales
  - Research Site, Eastbourne, Sussex
  - Research Site, Birmingham, West Midlands
  - Research Site, Bolton
  - Research Site, Bristol
  - Research Site, Cardiff
  - Research Site, Cleveland
  - Research Site, Edinburgh
  - Research Site, Falkirk
  - Research Site, Hull
  - Research Site, Kent
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Plymouth
  - Research Site, Sheffield
  - Research Site, Shrewsbury

REFERENCES:
- [Derived] Iversen P, McLeod DG, See WA, Morris T, Armstrong J, Wirth MP; Casodex Early Prostate Cancer Trialists' Group. Antiandrogen monotherapy in patients with localized or locally advanced prostate cancer: final results from the bicalutamide Early Prostate Cancer programme at a median follow-up of 9.7 years. BJU Int. 2010 Apr;105(8):1074-81. doi: 10.1111/j.1464-410X.2010.09319.x. PMID 22129214